CLINICAL TRIAL: NCT06829823
Title: Phase 2 Clinical Trial of Ablation Therapy With Intravesical N-803 In Combination With BCG or Gemcitabine in Participants With Intermediate-Risk Non-Muscle Invasive Papillary Bladder Cancer
Brief Title: Clinical Trial of Ablation Therapy in Participants With Intermediate-Risk Non-Muscle Invasive Papillary Bladder Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ResQ132A-NMIBC
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC)
Keywords: ResQ132A-NMIBC; Intermediate-Risk Non-Muscle Invasive Papillary Bladder Cancer; BCG; Gemcitabine; N-803
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — ALT-803; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-803 and BCG (Experimental): Combination treatment of 1) N-803 (400 μg): Weekly for 6 weeks (induction, re-induction); Monthly from month 3 through month 15 (maintenance) and 2) BCG (50mg): Weekly for 6 weeks (induction, re-induction)
  Interventions: Drug: N-803 and BCG
- N-803 and Gemcitabine (Experimental): Combination treatment of 1) N-803 (400 μg): Weekly for 6 weeks (induction, re-induction); Monthly from month 3 through month 15 (maintenance) and 2) Gemcitabine (2000mg): Weekly for 6 weeks (induction, re-induction)
  Interventions: Drug: N-803 and Gemcitabine

INTERVENTIONS:
Drug: N-803 and BCG — Combination therapy N-803 plus BCG
  Other Names: BCG; N-803; Bacillus Calmette-Guérin
  Arms: N-803 and BCG
Drug: N-803 and Gemcitabine — Combination therapy N-803 plus Gemcitabine
  Other Names: N-803; Gemcitabine; Gemzar
  Arms: N-803 and Gemcitabine

SUMMARY:
This is an open-label, phase 2, randomized study of intravesical N-803 plus BCG (experimental arm A) and intravesical N-803 plus gemcitabine (experimental arm B) in participants who have intermediate-risk Ta/T1 papillary disease. The primary objective of this study is to evaluate the efficacy of these experimental therapies without the need for surgical intervention by CR rate at month 3 or month 6 (for re-inducted participants).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Low-grade (LG) Ta papillary disease as determined by Investigator.
* History of LG NMIBC requiring treatment with transurethral resection of bladder tumors (TURBT). Note: This refers to a previous episode(s) and not to the current episode for which the participant is being screened. Any presence of variant histology, or LVI should be deemed high-risk.
* Negative voiding cytology for HG disease within 12 weeks prior to screening.
* Intermediate-risk disease, defined as having 1 or 2 of the following:

  1. Presence of >1 and < 5 tumors;
  2. Solitary tumor < 3 cm;
  3. Early or frequent recurrence (≥ 1 occurrence of LG NMIBC within 1 year of the current diagnosis at the initial screening visit).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2.
* Voluntary written informed consent and HIPAA authorization and agreement to comply with all protocol-specified procedures and follow-up evaluations.

Exclusion Criteria:

* Received BCG treatment for urothelial carcinoma.
* History of HG bladder cancer (papillary or CIS) in the past 2 years.
* Clinically significant urethral stricture that would preclude passage of a urethral catheter.
* Life expectancy < 2 years.
* Any of the following clinical laboratory values at the time of enrollment:

  1. Absolute lymphocyte count (ALC) > institutional lower limit of normal (LLN)
  2. Absolute neutrophil count (ANC) < 800/μL
  3. Platelets < 50,000/μL
  4. Aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) > 2 × upper limit of normal (ULN).
  5. Creatinine level > 3 × ULN. Note: Each study site should use its institutional LLN/ULN to determine eligibility.
* History of or evidence of muscle-invasive, locally advanced, metastatic and/or extravesical bladder cancer (inclusive of the prostatic urethra); or any other cancer within the past 5 years that is progressing or requires active treatment. Exceptions are adequately treated basal cell or squamous cell skin cancer that has undergone potentially curative therapy or in situ cervical cancer; adequately treated stage I or II cancer or stable prostate cancer from which the participant is currently in complete remission, and is under active surveillance or hormone control; or any other cancer that investigator feels is stable with permission of Medical Monitor.
* Suspicion of active upper tract urothelial malignancy.
* Currently receiving investigational or commercial anticancer agents or anticancer therapies other than BCG, N-803, and supportive care therapies for active disease.
* Symptomatic congestive heart failure (CHF), New York Heart Association (NYHA) Class III or IV heart failure, or other clinical signs of severe cardiac dysfunction.
* Severe/unstable angina pectoris, or myocardial infarction within 6 months prior to study entry.
* History or evidence of uncontrollable central nervous system [CNS] disease.
* Active systemic infection requiring parenteral antibiotic therapy. All prior infections must have resolved following optimal therapy.
* Concurrent febrile illness, active urinary tract infection, active tuberculosis, a history of hypotension or anaphylactic reactions.
* Ongoing chronic systemic steroid therapy required (>10 mg oral prednisone daily or equivalent).
* Women who are pregnant or nursing. Female participants of childbearing potential must have a negative pregnancy test and must adhere to using a medically acceptable method of birth control prior to screening and agree to continue its use during the study and for 7 months after the last dose of study drug, or be surgically sterilized (eg, hysterectomy or tubal ligation). Women of childbearing potential are defined as any female who has experienced menarche and who is NOT permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause. Males must agree to use barrier methods of birth control while on study and for 90 days post last dose of study drug.
* Other illness or condition, including laboratory abnormalities, which in the opinion of the Investigator would exclude the participant from participating in this study. This includes, but is not limited to, serious medical conditions or psychiatric illness likely to interfere with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Arms A and B at Month 3 and Month 6 | At Month 3 and Month 6
  Evaluate efficacy of experimental therapies with a) intravesical N-803 plus BCG or b) intravesical N-803 plus gemcitabine by CR rate at month 3 or month 6 (for re-inducted participants) in participants with intermediate-risk NMIBC.

SECONDARY OUTCOMES:
Efficacy of Arms A and B at by CR rate at each response assessment | At Month 3 through Month 36
  Evaluate efficacy of experimental therapy by CR rate at each response assessment.

IPD SHARING:
Plan to Share IPD: No